CLINICAL TRIAL: NCT00053937
Title: Phase I Trial Of Pirfenidone In Children With Neurofibromatosis Type 1 And Plexiform Neurofibromas
Brief Title: Pirfenidone in Treating Young Patients With Neurofibromatosis Type 1 and Plexiform Neurofibromas
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Prevention
Other Study IDs: CDR0000269598; NCI-03-C-0058A; NCT00050453 (obsolete NCT alias)
Record Dates: First submitted 2003-02-05; First posted 2003-02-06 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2004-04

CONDITIONS: Neurofibromatosis Type 1; Precancerous Condition
Keywords: plexiform neurofibroma; neurofibromatosis type 1
MeSH Terms: conditions — Neurofibromatosis 1; Precancerous Conditions; Neurofibroma, Plexiform | interventions — pirfenidone

INTERVENTIONS:
Drug: pirfenidone

SUMMARY:
RATIONALE: Chemoprevention therapy is the use of certain drugs to try to prevent the development or recurrence of cancer. Pirfenidone may slow the growth or prevent further development of plexiform neurofibromas.

PURPOSE: Phase I trial to study the effectiveness of pirfenidone in treating young patients who have neurofibromatosis type 1 and plexiform neurofibroma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the maximum tolerated dose or "comparable dose" of pirfenidone in pediatric patients with neurofibromatosis type 1 and inoperable, symptomatic plexiform neurofibromas.
* Determine the toxic effects of this drug in these patients.
* Determine the plasma pharmacokinetics of this drug in these patients.
* Determine, preliminarily, if this drug could be beneficial for pediatric patients with refractory solid tumors.
* Assess the quality of life of patients treated with this drug.

OUTLINE: This is an open-label, multicenter, dose-escalation study.

Patients receive oral pirfenidone three times daily on days 1-28. Courses repeat every 28 days for up to 2 years in the absence of disease progression or unacceptable toxicity.

Cohorts of 3-6 patients receive escalating doses of pirfenidone until the maximum tolerated dose (MTD) is determined. The MTD is defined as the dose preceding that at which 2 of 3 or 2 of 6 patients experience dose-limiting toxicity.

Quality of life is assessed at baseline, before course 4, and then after every 6 courses.

PROJECTED ACCRUAL: A total of 3-18 patients will be accrued for this study within 18 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of neurofibromatosis type 1 (NF1) AND
* Plexiform neurofibromas

  * Neurofibromas that have grown along the length of a nerve and may involve multiple fascicles and branches (spinal neurofibromas involve 2 or more levels with connection between the levels or extending laterally along the nerve)
  * Potential to cause significant morbidity such as:

    * Head and neck lesions that could compromise airway or great vessels
    * Brachial or lumbar plexus lesions that could cause nerve compression and loss of function
    * Lesions that could result in major deformity (e.g., orbital lesions) or significant cosmetic problems
    * Lesions of the extremity that cause limb hypertrophy or loss of function
    * Painful lesions
* Meets at least 1 other diagnostic criteria for NF1

  * 6 or more cafe-au-lait spots (at least 0.5 cm in prepubertal patients or at least 1.5 cm in postpubertal patients)
  * Freckling in the axilla or groin
  * Optic glioma
  * 2 or more Lisch nodules
  * Distinctive bony lesion (dysplasia of the sphenoid bone or dysplasia or thinning of long bone cortex)
  * First-degree relative with NF1
* Measurable plexiform neurofibromas

  * At least 3 cm in 1 dimension
  * Tumor resection not feasible
* No history of malignant peripheral nerve sheath tumor or other cancer
* No evidence of an active optic glioma requiring chemotherapy or radiotherapy
* No malignant glioma

PATIENT CHARACTERISTICS:

Age

* 3 to 21

Performance status

* Karnofsky 50-100% (over 10 years of age)
* Lansky 50-100% (10 years and under)

Life expectancy

* Not specified

Hematopoietic

* Absolute granulocyte count at least 1,500/mm^3
* Hemoglobin at least 9.0 g/dL
* Platelet count at least 150,000/mm^3

Hepatic

* Bilirubin normal
* SGPT no greater than 2 times upper limit of normal
* No clinically significant hepatic dysfunction that would preclude study participation

Renal

* Creatinine normal for age OR
* Creatinine clearance at least 70 mL/min

Cardiovascular

* No clinically significant cardiac dysfunction that would preclude study participation

Pulmonary

* No clinically significant pulmonary dysfunction that would preclude study participation

Other

* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 2 months after study
* Must be able to take pirfenidone orally
* No serious infections
* No clinically significant unrelated systemic illness or organ dysfunction that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* At least 30 days since prior immunotherapy
* No concurrent immunotherapy
* No concurrent hematopoietic growth factors

Chemotherapy

* At least 30 days since prior chemotherapy
* No concurrent chemotherapy directed at the tumor

Endocrine therapy

* At least 30 days since prior hormonal therapy directed at the tumor
* No concurrent hormonal therapy directed at the tumor

Radiotherapy

* At least 90 days since prior radiotherapy to the site of the plexiform neurofibroma
* No concurrent radiotherapy directed at the tumor

Surgery

* Not specified

Other

* Recovered from prior therapy
* More than 30 days since prior investigational agents
* No prior pirfenidone
* No other concurrent investigational agents

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Dates: Start 2002-12

CONTACTS AND LOCATIONS:
Overall Officials: Brigitte C. Widemann, MD, Study Chair — National Cancer Institute (NCI)
Locations (15):
- United States (15):
  - University of Alabama at Birmingham Comprehensive Cancer Center, Birmingham, Alabama
  - Children's National Medical Center, Washington D.C., District of Columbia
  - Children's Memorial Hospital - Chicago, Chicago, Illinois
  - Sidney Kimmel Comprehensive Cancer Center at Johns Hopkins, Baltimore, Maryland
  - Warren Grant Magnuson Clinical Center - NCI Clinical Studies Support, Bethesda, Maryland
  - Dana-Farber/Harvard Cancer Center at Dana Farber Cancer Institute, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Washington University School of Medicine, St Louis, Missouri
  - Beth Israel Medical Center - Singer Division, New York, New York
  - University Hospital at State University of New York - Upstate Medical University, Syracuse, New York
  - Cleveland Clinic Taussig Cancer Center, Cleveland, Ohio
  - Cancer Institute at Oregon Health and Science University, Portland, Oregon
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Children's Hospital of Pittsburgh, Pittsburgh, Pennsylvania
  - Texas Children's Cancer Center, Houston, Texas